CLINICAL TRIAL: NCT07196241
Title: Comprehensive Care for AYA: Needs Assessment Survey
Status: Not yet recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00136539; ONC-CCS-2505 (Other: Atrium Health Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Young Adult Cancer; Adolescent Cancer
Keywords: Adolescent; Young Adult; Cancer; AYA; Questionnaire; Needs assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and Young Adults with cancer: Participants diagnosed with cancer between the ages of 15-39 who have received or are receiving cancer-directed treatment at one of the participating centers per self-report.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — Questionnaires regarding cancer treatment and follow-up care, fertility preservation, clinical trial participation, general information (education on health- related topics, gender, and sexual orientation, perceived needs for resources, support areas, programs and activities.), emotional health and interpersonal relationships, financial burden and mental health status.

SUMMARY:
The goal of this observational study is to assess gaps in education about exercise, sexual health, fertility, survivorship, financial issues, interpersonal relationships, and clinical trial participation among adolescents and young adults with cancer.

Participants will be asked to complete a series of questionnaires.

DETAILED DESCRIPTION:
This descriptive study aims to assess current needs of adolescents and young adults with cancer.

Participants who were diagnosed with cancer between the ages of of 15-39 will be asked to complete questionnaires to provide information on their cancer treatments and follow-up care, fertility preservation, clinical trial participation, emotional health and interpersonal relationships, financial burden, mental health and additional general information (health related, sexual orientation, perceived needs for support, resources, programs and activities).

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with cancer between the ages of 15-39 per self-report. Participants may be enrolled at any age provided diagnosis was between ages 15-39.
* Individuals who have received or are receiving cancer-directed treatment (chemotherapy, immunotherapy, surgery and/or radiation) at one of the participating centers per self-report.

Exclusion Criteria:

* Severe emotional distress or anxiety that would limit compliance with study requirements per self-report.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants diagnosed with cancer between the ages of 15 and 39 and who received or are receiving treatment for their cancer at one of the centers participating in this research study.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Deficits in Education | At study enrollment
  The general information survey collects data on participants surrounding education on health-related topics, gender, and sexual orientation, as well as perceived needs for resources, support areas, programs and activities. The general information survey contains 12 items.
  There is no formal statistical analysis to be performed only summary statistics on completed survey items for observation thus there is no scoring needed or range of scores. Results will be observed using descriptive statistics. Due to the categorical nature of all variables, results will be reported in frequencies and percentages.
Preferred Format for Education | At study enrollment
  The General Information Survey collects data on participants surrounding education on health-related topics, gender, and sexual orientation, as well as perceived needs for resources, support areas, programs and activities. The general information survey contains 12 items.
  There is no formal statistical analysis to be performed only summary statistics on completed survey items for observation thus there is no scoring needed or range of scores. Results will be observed using descriptive statistics. Due to the categorical nature of all variables, results will be reported in frequencies and percentages.

OTHER OUTCOMES:
Deficit in Education by Covariates | At study enrollment
  Data on covariates will be collected with the Patient Demographic Information survey, Cancer History survey, Treatment Status and Follow-up Care survey, Fertility Preservation survey , Emotional Health and Interpersonal Relationships survey, Financial Burden survey and the Clinical Trial Participation Questionnaire.
  There is no formal statistical analysis to be performed only summary statistics on completed survey items for observation thus there is no scoring needed or range of scores. Results will be observed using cross tabulations reported in frequencies and percentages.
Focus Group Interest | At study enrollment
  Patients interested in serving on the AYA focus group will be identified using the single-item Interest in Focus Group Survey to provide contact information for a future focus group outside of this study.
  Results will be reported as binary (yes/no) for participation in the focus group via frequency and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Wofford, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No